CLINICAL TRIAL: NCT06319014
Title: Physical Activity to Mitigate PreEclampsia Risk (PAMPER)
Brief Title: Physical Activity to Mitigate PreEclampsia Risk
Acronym: PAMPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Linda May, Principal Investigator, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-001568
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Pregnant women will be randomized to one of four groups: aerobic exercise, resistance exercise, combination (aerobic + resistance), or control (no exercise). All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, rating of perceived exertion (RPE), 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AE Group (Experimental): The AE group will exercise on aerobic machines (i.e. treadmill, elliptical, bicycle)
  All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  Interventions: Behavioral: Exercise Modes
- RE Group (Experimental): The RE group will perform 12-15 repetitions of 10-12 resistance exercises in a circuit, for 3 sets, with a rest period of 30-60 seconds between sets as needed.[172] Seated isokinetic exercise using resistance machines will target all major muscle groups. Light dumbbells and resistance bands will be used if the participant is unable to lift the minimal load on machines. Core exercises will be performed at the end of the session (i.e. seated side bends)
  All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  Interventions: Behavioral: Exercise Modes
- AERE Group (Experimental): AERE group will alternate between AE exercise and RE; for this group, RE exercises will consist of 1 set of 12-15 repetitions of 4 resistance exercises, then 5 minutes of AE, then repeat this cycle with different exercises.
  All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  Interventions: Behavioral: Exercise Modes
- Control (No Intervention): The Control group will participate in weekly sessions that focus on stretching, breathing, and healthy lifestyle.

INTERVENTIONS:
Behavioral: Exercise Modes — Moderate intensity aerobic exercise Moderate intensity resistance exercise Moderate intensity combination exercise
  Arms: AE Group; AERE Group; RE Group

SUMMARY:
The purpose of this study is to compare the effects of aerobic (AE), resistance (RE), and combination (AERE) exercise throughout pregnancy on selected maternal and fetal/neonatal physiological variables in women at-risk for preeclampsia. The central hypothesis of this project is that exercise will decrease severity and occurrence of preeclampsia symptoms, thus improving maternal, pregnancy, and birth outcomes.

Aim 1. Determine the influence of different exercise modes during pregnancy at risk of preeclampsia on maternal cardiometabolic health.

Aim 2. Determine the most effective exercise mode in pregnancy at risk of preeclampsia on improving birth and infant health outcomes.

DETAILED DESCRIPTION:
Approximately 5% of pregnancies worldwide and in the United States were complicated by preeclampsia. Women who develop Preeclampsia in Pregnancy go on to develop Cardiovascular issues (Catov and other studies). Further, infants from preeclamptic pregnancies are at increased risk of mortality and co-morbid conditions (hypertension, excessive weight gain, increased BMI). However, preliminary data suggests that exercise will attenuate or prevent the severity and risk of preeclampsia; thus improving health for women and children. The purpose of this study is to compare the effects of aerobic (AE), resistance (RE), and combination (AERE) exercise throughout pregnancy on selected maternal and fetal/neonatal physiological variables in women at-risk for preeclampsia. The investigators hypothesize that following changes will occur:(1) improvements in the measurements of maternal resting heart rate, blood pressure, cardiometabolic risk (CMR) score, placental growth factor (PlGF), preeclampsia severity, onset of preeclampsia of symptoms at each time point (once per visit); and (2) improvements in birth and infant measurements of decreased C-sections, preterm deliveries, hospital stay, birth weight, placental efficiency at birth when exposed to different modes of maternal exercise compared no exercise (usual care) with greatest differences in AERE trained group. Ultimately, our goal is to determine which exercise program is most effective at attenuating or preventing preeclampsia and thus improving health outcomes for mother and child.

ELIGIBILITY:
Inclusion Criteria:

* healthy women, age 18-40 years, <16 weeks' gestation, with singleton pregnancy; women (BMI:18.5-45.0), sedentary, cleared by their obstetric provider.

Exclusion Criteria:

* pre-existing chronic conditions such as HIV, lupus, etc.; taking medicines that affect fetal development; and/or lack of telephone or email contact information).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (16wks) | 16 weeks gestation
  resting SBP
Systolic Blood Pressure (20wks) | 20 weeks gestation
  resting SBP
Systolic Blood Pressure (24wks) | 24 weeks gestation
  resting SBP
Systolic Blood Pressure (28wks) | 28 weeks gestation
  resting SBP
Systolic Blood Pressure (32wks) | 32 weeks gestation
  resting SBP
Systolic Blood Pressure (36wks) | 36 weeks gestation
  resting SBP
Maternal Cardiometabolic Risk (CMR) Score | during pregnancy
  summation of age- and sexstandardized z-scores for waist circumference (or BMI), triglycerides, systolic blood pressure (SBP), glucose (insulin or HOMA-IR), and inverse HDL, with a lower CMR score indicating lower risk
Symptom Occurrence | at delivery
  maternal medical record and questionnaire data for occurrence, signs, and symptoms of hypertension/pre-eclampsia
Placental Efficiency | at delivery
  placental weight gain and birth weight will be used to calculate placental efficiency
Birth Weight | at delivery
  infant birth weight
Infant Cardiometabolic Risk (CMR) Score | at delivery
  The CMR score will be a summation of age- and sex-standardized z-scores for abdominal circumference (or BMI),systolic blood pressure (SBP), glucose, and inverse HDL, with a lower CMR score indicating lower risk.

SECONDARY OUTCOMES:
Maternal Heart Rate (16wks) | 16 weeks gestation
  resting heart rate
Maternal Heart Rate (20wks) | 20 weeks gestation
  resting heart rate
Maternal Heart Rate (24wks) | 24 weeks gestation
  resting heart rate
Maternal Heart Rate (28wks) | 28 weeks gestation
  resting heart rate
Maternal Heart Rate (32wks) | 32 weeks gestation
  resting heart rate
Maternal Heart Rate (36wks) | 36 weeks gestation
  resting heart rate
Maternal Blood Pressure (16wks) | 16 weeks gestation
  resting bp
Maternal Blood Pressure (20wks) | 20 weeks gestation
  resting bp
Maternal Blood Pressure (24wks) | 24 weeks gestation
  resting bp
Maternal Blood Pressure (28wks) | 28 weeks gestation
  resting bp
Maternal Blood Pressure (32wks) | 32 weeks gestation
  resting bp
Maternal Blood Pressure (36wks) | 36 weeks gestation
  resting bp
Maternal Body Fat % (16wks) | 16 weeks gestation
  estimated body fat %
Maternal Body Fat % (20wks) | 20 weeks gestation
  estimated body fat %
Maternal Body Fat % (24wks) | 24 weeks gestation
  estimated body fat %
Maternal Body Fat % (28wks) | 28 weeks gestation
  estimated body fat %
Maternal Body Fat % (32wks) | 32 weeks gestation
  estimated body fat %
Maternal Body Fat % (36wks) | 36 weeks gestation
  estimated body fat %
Maternal Circumferences (16wks) | 16 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Maternal Circumferences (20wks) | 20 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Maternal Circumferences (24wks) | 24 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Maternal Circumferences (28wks) | 28 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Maternal Circumferences (32wks) | 32 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Maternal Circumferences (36wks) | 36 weeks gestation
  measurements will be assessed using a 3D Scanner and Gulick measuring tape
Gestational Weight Gain | at delivery
  weight at delivery minus pre-pregnancy weight
Delivery Mode | at delivery
  mode of delivery (i.e. vaginal, C-section, instrumentation) will be taken from EHR
Maternal Blood Glucose (16wks) | 16 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Glucose (20wks) | 20 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Glucose (24wks) | 24 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Glucose (28wks) | 28 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Glucose (32wks) | 32 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Glucose (36wks) | 36 weeks gestation
  blood glucose measured from venipuncture
Maternal Blood Lipids (16wks) | 16 weeks gestation
  blood lipids measured from venipuncture
Maternal Blood Lipids (20wks) | 20 weeks gestation
  blood lipids measured from venipuncture
Maternal Blood Lipids (24wks) | 24 weeks gestation
  blood lipids measured from venipuncture
Maternal Blood Lipids (28wks) | 28 weeks gestation
  blood lipids measured from venipuncture
Maternal Blood Lipids (32wks) | 32 weeks gestation
  blood lipids measured from venipuncture
Maternal Blood Lipids (36wks) | 36 weeks gestation
  blood lipids measured from venipuncture
Maternal Plasma Inflammatory Markers (16wks) | 16 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
Maternal Plasma Inflammatory Markers (20wks) | 20 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
Maternal Plasma Inflammatory Markers (24wks) | 24 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
Maternal Plasma Inflammatory Markers (28wks) | 28 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
Maternal Plasma Inflammatory Markers (32wks) | 32 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
Maternal Plasma Inflammatory Markers (36wks) | 36 weeks gestation
  inflammatory markers (i.e., IL-1b, IL-6, IL-8, TNF-a, CRP)
-omics Metabolites (16wks) | 16 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
-omics Metabolites (20wks) | 20 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
-omics Metabolites (24wks) | 24 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
-omics Metabolites (28wks) | 28 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
-omics Metabolites (32wks) | 32 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
-omics Metabolites (36wks) | 36 weeks gestation
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
Cord Blood and Placental Inflammatory Markers | at delivery
  inflammatory markers (i.e., IL-1b, IL-6, IL-8,TNF-a, CRP)
Cord Blood and Placental -omics Metabolites | at delivery
  MS core facility uses an Ultimate nano-liquid chromatography/Thermo Orbitrap Q-Exactive Plus and an Eskigent 425 micro-liquid chromatography/AB Sciex 5600+ Triple TOF (LC/MS) for our global proteomics and metabolomics analyses
Infant Body Morphometric Measures | at delivery
  circumferences and weight/length

CONTACTS AND LOCATIONS:
Overall Officials: Linda E May, MS, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data can be shared upon request to researchers